CLINICAL TRIAL: NCT01111240
Title: A Long Term Documentation to Demonstrate Long Term Efficacy and Safety of Humira® in Patients With Psoriatic Arthritis Under Conditions of Daily Practice
Brief Title: Efficacy and Safety of Humira® in Patients With Psoriatic Arthritis in Normal Medical Practice
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: HUM 05-3
Record Dates: First submitted 2010-02-26; First posted 2010-04-27 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Psoriatic Arthritis
Keywords: Humira; Long-term safety and effectiveness; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Psoriatic Arthritis: Participants with Psoriatic Arthritis prescribed adalimumab in routine clinical practice were observed from the first dose for up to 24 months.

SUMMARY:
This study is a documentation of effectiveness and safety of Humira in patients with psoriatic arthritis.

DETAILED DESCRIPTION:
Psoriatic Arthritis participants receiving adalimumab are evaluated in a prospective, non-interventional study (NIS) for 2 years. Patients receive adalimumab 40 mg every other week (eow), per its label. Efficacy and safety parameters are measured routinely at baseline and after 3, 6, 9, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion:

* 18 years of age or older (younger patients may be enrolled at the discretion of physician)
* Diagnosis of Psoriatic Arthritis (or any indication at the discretion of physician) and initiating adalimumab therapy
* Signed/dated Informed Consent

Exclusion:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical routine patients with psoriatic arthritis
Sampling Method: Non-Probability Sample
Enrollment: 4635 (Actual)
Dates: Start 2005-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bianca Wittig, MD, Study Director — Abbvie Deutschland GmbH & Co. KG, Medical Department
Locations (509):
- Germany (509):
  - Site Reference ID/Investigator# 35035, Aachen
  - Site Reference ID/Investigator# 64288, Aachen
  - Site Reference ID/Investigator# 35509, Ahlen
  - Site Reference ID/Investigator# 53118, Ahrensburg
  - Site Reference ID/Investigator# 35042, Altenburg
  - Site Reference ID/Investigator# 35045, Altenholz
  - Site Reference ID/Investigator# 35048, Amberg
  - Site Reference ID/Investigator# 96243, Annaberg-Buchholz
  - Site Reference ID/Investigator# 53205, Arnstadt
  - Site Reference ID/Investigator# 53091, Artern
  - Site Reference ID/Investigator# 33348, Augsburg
  - Site Reference ID/Investigator# 33357, Bad Abbach
  - Site Reference ID/Investigator# 35085, Bad Aibling
  - Site Reference ID/Investigator# 57895, Bad Aibling
  - Site Reference ID/Investigator# 91097, Bad Bentheim
  - Site Reference ID/Investigator# 35524, Bad Bentheim
  - Site Reference ID/Investigator# 35572, Bad Bramstedt
  - Site Reference ID/Investigator# 64304, Bad Bramstedt
  - Site Reference ID/Investigator# 33371, Bad Endbach
  - Site Reference ID/Investigator# 53278, Bad Endbach
  - Site Reference ID/Investigator# 91084, Bad Homburg
  - Site Reference ID/Investigator# 33377, Bad Iburg
  - Site Reference ID/Investigator# 33381, Bad Iburg
  - Site Reference ID/Investigator# 53068, Bad Kissingen
  - Site Reference ID/Investigator# 33386, Bad Kreuznach
  - Site Reference ID/Investigator# 35574, Bad Kreuznach
  - Site Reference ID/Investigator# 33390, Bad Liebenwerda
  - Site Reference ID/Investigator# 33395, Bad Münder am Deister
  - Site Reference ID/Investigator# 96245, Bad Münder am Deister
  - Site Reference ID/Investigator# 91094, Bad Nauheim
  - Site Reference ID/Investigator# 35577, Bad Neuenahr
  - Site Reference ID/Investigator# 53181, Bad Neuenahr
  - Site Reference ID/Investigator# 57885, Bad Oeynhausen
  - Site Reference ID/Investigator# 33403, Bad Rappenau
  - Site Reference ID/Investigator# 53060, Bad Salzungen
  - Site Reference ID/Investigator# 91079, Bad Salzungen
  - Site Reference ID/Investigator# 53254, Bad Schlema
  - Site Reference ID/Investigator# 33416, Bad Staffelstein
  - Site Reference ID/Investigator# 33420, Bad Sülze
  - Site Reference ID/Investigator# 57890, Bad Tölz
  - Site Reference ID/Investigator# 33424, Baden-Baden
  - Site Reference ID/Investigator# 33428, Bamberg
  - Site Reference ID/Investigator# 33434, Bautzen
  - Site Reference ID/Investigator# 33437, Bautzen
  - Site Reference ID/Investigator# 53231, Bayreuth
  - Site Reference ID/Investigator# 33441, Bayreuth
  - Site Reference ID/Investigator# 33445, Bayreuth
  - Site Reference ID/Investigator# 68595, Bergen
  - Site Reference ID/Investigator# 33459, Berlin
  - Site Reference ID/Investigator# 35087, Berlin
  - Site Reference ID/Investigator# 53058, Berlin
  - Site Reference ID/Investigator# 53241, Berlin
  - Site Reference ID/Investigator# 53242, Berlin
  - Site Reference ID/Investigator# 33647, Berlin
  - Site Reference ID/Investigator# 57909, Berlin
  - Site Reference ID/Investigator# 53061, Berlin
  - Site Reference ID/Investigator# 53059, Berlin
  - Site Reference ID/Investigator# 68842, Berlin
  - Site Reference ID/Investigator# 33657, Berlin
  - Site Reference ID/Investigator# 53105, Berlin
  - Site Reference ID/Investigator# 98535, Berlin
  - Site Reference ID/Investigator# 34245, Berlin
  - Site Reference ID/Investigator# 33682, Berlin
  - Site Reference ID/Investigator# 68594, Berlin
  - Site Reference ID/Investigator# 34268, Berlin
  - Site Reference ID/Investigator# 33654, Berlin
  - Site Reference ID/Investigator# 64284, Berlin
  - Site Reference ID/Investigator# 35596, Berlin
  - Site Reference ID/Investigator# 35600, Berlin
  - Site Reference ID/Investigator# 53081, Berlin
  - Site Reference ID/Investigator# 53244, Berlin
  - Site Reference ID/Investigator# 91075, Berlin
  - Site Reference ID/Investigator# 64287, Berlin
  - Site Reference ID/Investigator# 34261, Berlin
  - Site Reference ID/Investigator# 33686, Berlin
  - Site Reference ID/Investigator# 64286, Berlin
  - Site Reference ID/Investigator# 52990, Berlin
  - Site Reference ID/Investigator# 52995, Berlin
  - Site Reference ID/Investigator# 35549, Berlin
  - Site Reference ID/Investigator# 53090, Berlin
  - Site Reference ID/Investigator# 35553, Berlin
  - Site Reference ID/Investigator# 57893, Berlin-Weissensee
  - Site Reference ID/Investigator# 35555, Bernau
  - Site Reference ID/Investigator# 53213, Bernsbach
  - Site Reference ID/Investigator# 34274, Beverungen
  - Site Reference ID/Investigator# 53085, Bietigheim-Bissingen
  - Site Reference ID/Investigator# 53268, Bietigheim-Bissingen
  - Site Reference ID/Investigator# 34284, Blankenburg/Hart
  - Site Reference ID/Investigator# 34287, Blaubeuren Abbey
  - Site Reference ID/Investigator# 34290, Bocholt
  - Site Reference ID/Investigator# 35640, Bochum
  - Site Reference ID/Investigator# 53196, Bochum
  - Site Reference ID/Investigator# 53179, Bochum
  - Site Reference ID/Investigator# 57908, Bochum
  - Site Reference ID/Investigator# 35643, Bogen
  - Site Reference ID/Investigator# 34301, Bonn
  - Site Reference ID/Investigator# 34295, Bonn
  - Site Reference ID/Investigator# 34306, Braunschweig
  - Site Reference ID/Investigator# 53234, Breitenbrunn
  - Site Reference ID/Investigator# 35608, Bremen
  - Site Reference ID/Investigator# 52987, Bremen
  - Site Reference ID/Investigator# 53107, Bremen
  - Site Reference ID/Investigator# 53247, Bremen
  - Site Reference ID/Investigator# 91073, Bremerhaven
  - Site Reference ID/Investigator# 34265, Buch
  - Site Reference ID/Investigator# 64291, Buch
  - Site Reference ID/Investigator# 68584, Burgstädt
  - Site Reference ID/Investigator# 81599, Chemnitz
  - Site Reference ID/Investigator# 34698, Chemnitz
  - Site Reference ID/Investigator# 57902, Chemnitz
  - Site Reference ID/Investigator# 35094, Chemnitz
  - Site Reference ID/Investigator# 53262, Cologne
  - Site Reference ID/Investigator# 64298, Cologne
  - Site Reference ID/Investigator# 64293, Cologne
  - Site Reference ID/Investigator# 33988, Cologne
  - Site Reference ID/Investigator# 53193, Cologne
  - Site Reference ID/Investigator# 53071, Cologne
  - Site Reference ID/Investigator# 35236, Cologne
  - Site Reference ID/Investigator# 64300, Cologne
  - Site Reference ID/Investigator# 72857, Cologne
  - Site Reference ID/Investigator# 34710, Cottbus
  - Site Reference ID/Investigator# 53184, Cottbus
  - Site Reference ID/Investigator# 64303, Darmstadt
  - Site Reference ID/Investigator# 35620, Darmstadt
  - Site Reference ID/Investigator# 34724, Deggendorf
  - Site Reference ID/Investigator# 53209, Delmenhorst
  - Site Reference ID/Investigator# 53089, Delmenhorst
  - Site Reference ID/Investigator# 91077, Dinslaken
  - Site Reference ID/Investigator# 34741, Dortmund
  - Site Reference ID/Investigator# 35637, Dortmund
  - Site Reference ID/Investigator# 35633, Dortmund
  - Site Reference ID/Investigator# 57899, Dresden
  - Site Reference ID/Investigator# 35172, Dresden
  - Site Reference ID/Investigator# 34753, Dresden
  - Site Reference ID/Investigator# 53069, Dresden
  - Site Reference ID/Investigator# 34747, Dresden
  - Site Reference ID/Investigator# 34750, Dresden
  - Site Reference ID/Investigator# 34759, Dresden
  - Site Reference ID/Investigator# 68590, Dresden
  - Site Reference ID/Investigator# 53182, Dresden
  - Site Reference ID/Investigator# 91081, Dresden
  - Site Reference ID/Investigator# 68592, Dresden
  - Site Reference ID/Investigator# 57904, Dresden
  - Site Reference ID/Investigator# 34777, Duisburg
  - Site Reference ID/Investigator# 53072, Duisburg
  - Site Reference ID/Investigator# 98537, Duisburg
  - Site Reference ID/Investigator# 53266, Düren
  - Site Reference ID/Investigator# 34772, Düsseldorf
  - Site Reference ID/Investigator# 64302, Düsseldorf
  - Site Reference ID/Investigator# 34783, Eberswalde
  - Site Reference ID/Investigator# 53194, Eberswalde
  - Site Reference ID/Investigator# 53065, Eisenach
  - Site Reference ID/Investigator# 72856, Eisenach
  - Site Reference ID/Investigator# 53000, Eisleben Lutherstadt
  - Site Reference ID/Investigator# 35181, Elmshorn
  - Site Reference ID/Investigator# 53114, Eppstein
  - Site Reference ID/Investigator# 53221, Erftstadt
  - Site Reference ID/Investigator# 53070, Erfurt
  - Site Reference ID/Investigator# 53258, Erfurt
  - Site Reference ID/Investigator# 53259, Erfurt
  - Site Reference ID/Investigator# 57900, Erfurt
  - Site Reference ID/Investigator# 34808, Erfurt
  - Site Reference ID/Investigator# 35095, Erfurt
  - Site Reference ID/Investigator# 57901, Erkrath
  - Site Reference ID/Investigator# 34820, Erlangen
  - Site Reference ID/Investigator# 57896, Erlangen
  - Site Reference ID/Investigator# 35195, Essen
  - Site Reference ID/Investigator# 35198, Essen
  - Site Reference ID/Investigator# 53219, Esslingen am Neckar
  - Site Reference ID/Investigator# 35201, Feldafing
  - Site Reference ID/Investigator# 35204, Flensburg
  - Site Reference ID/Investigator# 34832, Forchheim
  - Site Reference ID/Investigator# 35209, Frankenberg
  - Site Reference ID/Investigator# 64283, Frankfurt
  - Site Reference ID/Investigator# 34839, Frankfurt
  - Site Reference ID/Investigator# 35212, Fraureuth
  - Site Reference ID/Investigator# 91078, Frechen
  - Site Reference ID/Investigator# 35218, Freiberg
  - Site Reference ID/Investigator# 34853, Freiburg im Breisgau
  - Site Reference ID/Investigator# 34856, Freiburg im Breisgau
  - Site Reference ID/Investigator# 34860, Freiburg im Breisgau
  - Site Reference ID/Investigator# 35100, Freystadt
  - Site Reference ID/Investigator# 35223, Friedrichroda
  - Site Reference ID/Investigator# 68843, Garching
  - Site Reference ID/Investigator# 34878, Gelsenkirchen
  - Site Reference ID/Investigator# 68591, Gelsenkirchen
  - Site Reference ID/Investigator# 34882, Gera
  - Site Reference ID/Investigator# 57907, Gera
  - Site Reference ID/Investigator# 64285, Gera
  - Site Reference ID/Investigator# 64294, Gera
  - Site Reference ID/Investigator# 57897, Gera
  - Site Reference ID/Investigator# 53222, Gera
  - Site Reference ID/Investigator# 34886, Giessen
  - Site Reference ID/Investigator# 53116, Gornau
  - Site Reference ID/Investigator# 34895, Goslar
  - Site Reference ID/Investigator# 68589, Gotha
  - Site Reference ID/Investigator# 52998, Göttingen
  - Site Reference ID/Investigator# 35493, Gräfelfing
  - Site Reference ID/Investigator# 53224, Greifswald
  - Site Reference ID/Investigator# 57889, Greifswald
  - Site Reference ID/Investigator# 64289, Greifswald
  - Site Reference ID/Investigator# 34903, Greifswald
  - Site Reference ID/Investigator# 58122, Greifswald
  - Site Reference ID/Investigator# 53106, Gronau
  - Site Reference ID/Investigator# 91070, Großenhain
  - Site Reference ID/Investigator# 34911, Güstrow
  - Site Reference ID/Investigator# 34936, Halle
  - Site Reference ID/Investigator# 34939, Halle
  - Site Reference ID/Investigator# 53067, Halle
  - Site Reference ID/Investigator# 53236, Halle
  - Site Reference ID/Investigator# 81601, Halle
  - Site Reference ID/Investigator# 34921, Halle
  - Site Reference ID/Investigator# 34943, Halle
  - Site Reference ID/Investigator# 34931, Halle
  - Site Reference ID/Investigator# 53063, Hamburg
  - Site Reference ID/Investigator# 53183, Hamburg
  - Site Reference ID/Investigator# 96237, Hamburg
  - Site Reference ID/Investigator# 34969, Hamburg
  - Site Reference ID/Investigator# 53073, Hamburg
  - Site Reference ID/Investigator# 34951, Hamburg
  - Site Reference ID/Investigator# 53276, Hamburg
  - Site Reference ID/Investigator# 34957, Hamburg
  - Site Reference ID/Investigator# 96242, Hamburg
  - Site Reference ID/Investigator# 35451, Hamburg
  - Site Reference ID/Investigator# 53198, Hamburg
  - Site Reference ID/Investigator# 35113, Hamburg
  - Site Reference ID/Investigator# 35006, Hamburg
  - Site Reference ID/Investigator# 53186, Hamburg
  - Site Reference ID/Investigator# 53212, Hamburg
  - Site Reference ID/Investigator# 53206, Hamburg
  - Site Reference ID/Investigator# 34960, Hamburg
  - Site Reference ID/Investigator# 53199, Hamburg
  - Site Reference ID/Investigator# 35448, Hamburg
  - Site Reference ID/Investigator# 34954, Hamburg
  - Site Reference ID/Investigator# 34997, Hamburg
  - Site Reference ID/Investigator# 34993, Hamburg
  - Site Reference ID/Investigator# 53098, Hamburg
  - Site Reference ID/Investigator# 53279, Hamburg
  - Site Reference ID/Investigator# 72854, Hamburg
  - Site Reference ID/Investigator# 34982, Hamburg
  - Site Reference ID/Investigator# 34985, Hamburg
  - Site Reference ID/Investigator# 35110, Hamburg
  - Site Reference ID/Investigator# 53066, Hamburg
  - Site Reference ID/Investigator# 53248, Hamburg
  - Site Reference ID/Investigator# 34973, Hamburg
  - Site Reference ID/Investigator# 35018, Hanau
  - Site Reference ID/Investigator# 33711, Hanover
  - Site Reference ID/Investigator# 53100, Hanover
  - Site Reference ID/Investigator# 68582, Hanover
  - Site Reference ID/Investigator# 53083, Hanover
  - Site Reference ID/Investigator# 64301, Hanover
  - Site Reference ID/Investigator# 53256, Harrislee
  - Site Reference ID/Investigator# 33797, Heidelberg
  - Site Reference ID/Investigator# 33804, Heidelberg
  - Site Reference ID/Investigator# 35118, Heidelberg
  - Site Reference ID/Investigator# 91083, Heidelberg
  - Site Reference ID/Investigator# 33800, Heidelberg
  - Site Reference ID/Investigator# 33807, Heidelberg
  - Site Reference ID/Investigator# 33817, Heilbad Heiligenstadt
  - Site Reference ID/Investigator# 53057, Heilbad Heiligenstadt
  - Site Reference ID/Investigator# 64297, Herne
  - Site Reference ID/Investigator# 57894, Herrsching am Ammersee
  - Site Reference ID/Investigator# 68586, Herten
  - Site Reference ID/Investigator# 53272, Hildburghausen
  - Site Reference ID/Investigator# 53080, Hilden
  - Site Reference ID/Investigator# 53097, Hildesheim
  - Site Reference ID/Investigator# 33833, Hof
  - Site Reference ID/Investigator# 33841, Hofheim
  - Site Reference ID/Investigator# 114015, Hohen Neuendorf
  - Site Reference ID/Investigator# 33844, Hohenfelde
  - Site Reference ID/Investigator# 53084, Holzkirchen
  - Site Reference ID/Investigator# 53092, Homburg
  - Site Reference ID/Investigator# 91085, Homburg
  - Site Reference ID/Investigator# 53109, Hoyerswerda
  - Site Reference ID/Investigator# 33857, Immenstadt im Allgäu
  - Site Reference ID/Investigator# 98538, Ingoldstadt
  - Site Reference ID/Investigator# 33934, Ingolstadt
  - Site Reference ID/Investigator# 53111, Ingolstadt
  - Site Reference ID/Investigator# 53053, Jena
  - Site Reference ID/Investigator# 53055, Jena
  - Site Reference ID/Investigator# 5305, Jena
  - Site Reference ID/Investigator# 33941, Jülich
  - Site Reference ID/Investigator# 33945, Kahla
  - Site Reference ID/Investigator# 35123, Kahla
  - Site Reference ID/Investigator# 33949, Kaiserslautern
  - Site Reference ID/Investigator# 52992, Kamenz
  - Site Reference ID/Investigator# 33960, Karlsruhe
  - Site Reference ID/Investigator# 35483, Karlstadt am Main
  - Site Reference ID/Investigator# 53192, Kassel
  - Site Reference ID/Investigator# 33963, Kassel
  - Site Reference ID/Investigator# 33967, Katzhütte
  - Site Reference ID/Investigator# 53229, Kiel
  - Site Reference ID/Investigator# 72859, Kleinmachnow
  - Site Reference ID/Investigator# 53233, Koblenz
  - Site Reference ID/Investigator# 34001, Königs Wusterhausen
  - Site Reference ID/Investigator# 91076, Krefeld
  - Site Reference ID/Investigator# 91093, Krefeld
  - Site Reference ID/Investigator# 53108, Krefeld
  - Site Reference ID/Investigator# 34007, Kressbronn
  - Site Reference ID/Investigator# 34083, Kronach
  - Site Reference ID/Investigator# 53101, Kyritz
  - Site Reference ID/Investigator# 34004, Lahr
  - Site Reference ID/Investigator# 35244, Landau
  - Site Reference ID/Investigator# 64290, Langenfeld
  - Site Reference ID/Investigator# 53245, Leinefelde
  - Site Reference ID/Investigator# 53115, Leipzig
  - Site Reference ID/Investigator# 53087, Leipzig
  - Site Reference ID/Investigator# 34105, Leipzig
  - Site Reference ID/Investigator# 34108, Leipzig
  - Site Reference ID/Investigator# 53197, Leipzig
  - Site Reference ID/Investigator# 53052, Leipzig
  - Site Reference ID/Investigator# 53211, Leipzig
  - Site Reference ID/Investigator# 53088, Leverkusen
  - Site Reference ID/Investigator# 34122, Lichtenstein
  - Site Reference ID/Investigator# 53180, Lingen
  - Site Reference ID/Investigator# 35253, Lippstadt
  - Site Reference ID/Investigator# 96240, Löbau
  - Site Reference ID/Investigator# 35259, Ludwigsfelde
  - Site Reference ID/Investigator# 53195, Ludwigshafen
  - Site Reference ID/Investigator# 53249, Ludwigslust
  - Site Reference ID/Investigator# 53110, Lübeck
  - Site Reference ID/Investigator# 34135, Lübeck
  - Site Reference ID/Investigator# 53074, Lüdenscheid
  - Site Reference ID/Investigator# 96239, Lüneburg
  - Site Reference ID/Investigator# 34146, Magdeburg
  - Site Reference ID/Investigator# 34149, Magdeburg
  - Site Reference ID/Investigator# 91082, Magdeburg
  - Site Reference ID/Investigator# 64292, Magdeburg
  - Site Reference ID/Investigator# 68583, Magdeburg
  - Site Reference ID/Investigator# 53230, Magdeburg
  - Site Reference ID/Investigator# 64305, Magdeburg
  - Site Reference ID/Investigator# 53075, Mainz
  - Site Reference ID/Investigator# 68593, Mainz
  - Site Reference ID/Investigator# 34179, Mannheim
  - Site Reference ID/Investigator# 34191, Marktredwitz
  - Site Reference ID/Investigator# 34195, Marl
  - Site Reference ID/Investigator# 34199, Meissen
  - Site Reference ID/Investigator# 53269, Melsungen
  - Site Reference ID/Investigator# 53078, Memmingen
  - Site Reference ID/Investigator# 35284, Menz
  - Site Reference ID/Investigator# 35286, Minden
  - Site Reference ID/Investigator# 34207, Mittelherwigsdorf
  - Site Reference ID/Investigator# 57883, Moenkeburg
  - Site Reference ID/Investigator# 34217, Mönchengladbach
  - Site Reference ID/Investigator# 34212, Mönchengladbach
  - Site Reference ID/Investigator# 53095, Mönchengladbach
  - Site Reference ID/Investigator# 53261, Mönchengladbach
  - Site Reference ID/Investigator# 64282, Munich
  - Site Reference ID/Investigator# 34039, Munich
  - Site Reference ID/Investigator# 57892, Munich
  - Site Reference ID/Investigator# 64295, Munich
  - Site Reference ID/Investigator# 35294, Munich
  - Site Reference ID/Investigator# 34234, Munich
  - Site Reference ID/Investigator# 91080, Munich
  - Site Reference ID/Investigator# 34042, Munich
  - Site Reference ID/Investigator# 53270, Munich
  - Site Reference ID/Investigator# 34223, Mühlhausen
  - Site Reference ID/Investigator# 35291, Mülheim
  - Site Reference ID/Investigator# 53235, Mülheim
  - Site Reference ID/Investigator# 34228, Müllheim
  - Site Reference ID/Investigator# 53062, Münster
  - Site Reference ID/Investigator# 68587, Münster
  - Site Reference ID/Investigator# 34047, Münster
  - Site Reference ID/Investigator# 53093, Münster
  - Site Reference ID/Investigator# 91096, Münster
  - Site Reference ID/Investigator# 53246, Naila
  - Site Reference ID/Investigator# 53271, Nastätten
  - Site Reference ID/Investigator# 35305, Naumburg
  - Site Reference ID/Investigator# 34051, Naunhof
  - Site Reference ID/Investigator# 34060, Neubrandenburg
  - Site Reference ID/Investigator# 34063, Neuburg am Inn
  - Site Reference ID/Investigator# 53220, Neunkirchen
  - Site Reference ID/Investigator# 35312, Neuss
  - Site Reference ID/Investigator# 34075, Neustadt
  - Site Reference ID/Investigator# 34079, Niefern-Öschelbronn
  - Site Reference ID/Investigator# 34157, Nienburg
  - Site Reference ID/Investigator# 57891, Nienburg
  - Site Reference ID/Investigator# 52997, Nordhausen
  - Site Reference ID/Investigator# 52999, Nordhausen
  - Site Reference ID/Investigator# 53277, Nordhausen
  - Site Reference ID/Investigator# 53054, Nuremberg
  - Site Reference ID/Investigator# 68588, Nuremberg
  - Site Reference ID/Investigator# 53112, Nuremberg
  - Site Reference ID/Investigator# 96244, Oberhausen
  - Site Reference ID/Investigator# 34172, Oelsnitz
  - Site Reference ID/Investigator# 53104, Oelsnitz
  - Site Reference ID/Investigator# 34175, Offenburg
  - Site Reference ID/Investigator# 33491, Oldenburg
  - Site Reference ID/Investigator# 57886, Oldenburg
  - Site Reference ID/Investigator# 91067, Oschatz
  - Site Reference ID/Investigator# 53207, Osnabrück
  - Site Reference ID/Investigator# 81600, Osnabrück
  - Site Reference ID/Investigator# 53228, Ostseebad Damp
  - Site Reference ID/Investigator# 35334, Paderborn
  - Site Reference ID/Investigator# 33507, Parchim
  - Site Reference ID/Investigator# 35339, Passau
  - Site Reference ID/Investigator# 72858, Peitz
  - Site Reference ID/Investigator# 53096, Petershagen
  - Site Reference ID/Investigator# 53086, Pinneberg
  - Site Reference ID/Investigator# 53232, Pirna
  - Site Reference ID/Investigator# 33522, Planegg
  - Site Reference ID/Investigator# 33527, Plauen
  - Site Reference ID/Investigator# 96278, Plochingen
  - Site Reference ID/Investigator# 33469, Potsdam
  - Site Reference ID/Investigator# 33465, Potsdam
  - Site Reference ID/Investigator# 96236, Potsdam
  - Site Reference ID/Investigator# 53281, Potsdam
  - Site Reference ID/Investigator# 33475, Prüm
  - Site Reference ID/Investigator# 33478, Püttlingen
  - Site Reference ID/Investigator# 53257, Püttlingen
  - Site Reference ID/Investigator# 91120, Püttlingen
  - Site Reference ID/Investigator# 53094, Quedlinburg
  - Site Reference ID/Investigator# 53265, Querfurt
  - Site Reference ID/Investigator# 33483, Radebeul
  - Site Reference ID/Investigator# 35346, Radebeul
  - Site Reference ID/Investigator# 53280, Ratingen
  - Site Reference ID/Investigator# 57888, Ratingen
  - Site Reference ID/Investigator# 33487, Ratzeburg
  - Site Reference ID/Investigator# 33889, Regensburg
  - Site Reference ID/Investigator# 57912, Regensburg
  - Site Reference ID/Investigator# 57911, Regensburg
  - Site Reference ID/Investigator# 53264, Regensburg
  - Site Reference ID/Investigator# 33901, Rendsburg
  - Site Reference ID/Investigator# 52991, Ribnitz-Damgarten
  - Site Reference ID/Investigator# 53267, Riesa
  - Site Reference ID/Investigator# 33910, Riesa
  - Site Reference ID/Investigator# 33913, Rinteln
  - Site Reference ID/Investigator# 33922, Rostock
  - Site Reference ID/Investigator# 33926, Rostock
  - Site Reference ID/Investigator# 33930, Rothenburg
  - Site Reference ID/Investigator# 53113, Rudolstadt
  - Site Reference ID/Investigator# 35361, Rüdersdorf
  - Site Reference ID/Investigator# 34015, Saarbrücken
  - Site Reference ID/Investigator# 91071, Saarlouis
  - Site Reference ID/Investigator# 35382, Saint Martin
  - Site Reference ID/Investigator# 34022, Salzwedel
  - Site Reference ID/Investigator# 34026, Sande
  - Site Reference ID/Investigator# 53208, Schleiz
  - Site Reference ID/Investigator# 91074, Schlettau
  - Site Reference ID/Investigator# 33533, Schneeberg
  - Site Reference ID/Investigator# 33538, Schramberg
  - Site Reference ID/Investigator# 33541, Schutterwald
  - Site Reference ID/Investigator# 35370, Schwandorf in Bayern
  - Site Reference ID/Investigator# 91072, Schwandorf in Bayern
  - Site Reference ID/Investigator# 57905, Schwedt
  - Site Reference ID/Investigator# 72855, Schweina
  - Site Reference ID/Investigator# 33548, Schwerin
  - Site Reference ID/Investigator# 35375, Schwerin
  - Site Reference ID/Investigator# 33554, Schwerte
  - Site Reference ID/Investigator# 33558, Seesen
  - Site Reference ID/Investigator# 33566, Sinsheim
  - Site Reference ID/Investigator# 33571, Soltau
  - Site Reference ID/Investigator# 53255, Spelle
  - Site Reference ID/Investigator# 33584, Stadtbergen
  - Site Reference ID/Investigator# 98539, Stolberg
  - Site Reference ID/Investigator# 53218, Storkow
  - Site Reference ID/Investigator# 53082, Straubing
  - Site Reference ID/Investigator# 33603, Stuttgart
  - Site Reference ID/Investigator# 33606, Stuttgart
  - Site Reference ID/Investigator# 33610, Stuttgart
  - Site Reference ID/Investigator# 33597, Stuttgart
  - Site Reference ID/Investigator# 53210, Suhl
  - Site Reference ID/Investigator# 53223, Suhl
  - Site Reference ID/Investigator# 35388, Suhl
  - Site Reference ID/Investigator# 33624, Torgelow
  - Site Reference ID/Investigator# 53077, Treuenbrietzen
  - Site Reference ID/Investigator# 57906, Treuenbrietzen
  - Site Reference ID/Investigator# 53200, Tuttlingen
  - Site Reference ID/Investigator# 57910, Ueberlingen-Nussdorf
  - Site Reference ID/Investigator# 33640, Ulm
  - Site Reference ID/Investigator# 33723, Ulm
  - Site Reference ID/Investigator# 81602, Unna
  - Site Reference ID/Investigator# 96241, Varel
  - Site Reference ID/Investigator# 98536, Verden an der Aller
  - Site Reference ID/Investigator# 72860, Viersen
  - Site Reference ID/Investigator# 33736, Villingen-Schwenningen
  - Site Reference ID/Investigator# 33741, Waltrop
  - Site Reference ID/Investigator# 53243, Wannsee
  - Site Reference ID/Investigator# 72853, Wasserburg
  - Site Reference ID/Investigator# 33748, Weener
  - Site Reference ID/Investigator# 33851, Welzow
  - Site Reference ID/Investigator# 35407, Wiesbaden
  - Site Reference ID/Investigator# 33764, Wiesbaden
  - Site Reference ID/Investigator# 52989, Wiesbaden
  - Site Reference ID/Investigator# 33771, Wilhelmshaven
  - Site Reference ID/Investigator# 53076, Winsen
  - Site Reference ID/Investigator# 33775, Wismar
  - Site Reference ID/Investigator# 33779, Wittlich
  - Site Reference ID/Investigator# 91095, Wittmund
  - Site Reference ID/Investigator# 96235, Wolfenbüttel
  - Site Reference ID/Investigator# 91068, Wuppertal
  - Site Reference ID/Investigator# 91069, Wuppertal
  - Site Reference ID/Investigator# 35419, Wuppertal
  - Site Reference ID/Investigator# 57884, Wurzen
  - Site Reference ID/Investigator# 33717, Würzburg
  - Site Reference ID/Investigator# 57903, Würzburg
  - Site Reference ID/Investigator# 53064, Zeitz
  - Site Reference ID/Investigator# 33863, Zerbst
  - Site Reference ID/Investigator# 33866, Zeven
  - Site Reference ID/Investigator# 64299, Zschopau
  - Site Reference ID/Investigator# 52996, Zwickau
  - Site Reference ID/Investigator# 33875, Zwickau
  - Site Reference ID/Investigator# 52993, Zwickau
  - Site Reference ID/Investigator# 53056, Zwickau
  - Site Reference ID/Investigator# 53102, Zwickau
  - Site Reference ID/Investigator# 52994, Zwickau
  - Site Reference ID/Investigator# 53226, Zwickau
  - Site Reference ID/Investigator# 53260, Zwickau
  - Site Reference ID/Investigator# 33879, Zwiesel

REFERENCES:
- [Derived] Behrens F, Koehm M, Schwaneck EC, Schmalzing M, Wittig BM, Gnann H, Greger G, Tony HP, Burkhardt H. Addition or removal of concomitant methotrexate alters adalimumab effectiveness in rheumatoid arthritis but not psoriatic arthritis. Scand J Rheumatol. 2019 Sep;48(5):375-382. doi: 10.1080/03009742.2019.1600717. Epub 2019 Jul 16. PMID 31311386
- [Derived] Behrens F, Koehm M, Schwaneck EC, Schmalzing M, Gnann H, Greger G, Tony HP, Burkhardt H. Minimal disease activity is a stable measure of therapeutic response in psoriatic arthritis patients receiving treatment with adalimumab. Rheumatology (Oxford). 2018 Nov 1;57(11):1938-1946. doi: 10.1093/rheumatology/key203. PMID 30010891
- [Derived] Behrens F, Koehm M, Thaci D, Gnann H, Greger G, Maria Wittig B, Burkhardt H. Anti-citrullinated protein antibodies are linked to erosive disease in an observational study of patients with psoriatic arthritis. Rheumatology (Oxford). 2016 Oct;55(10):1791-5. doi: 10.1093/rheumatology/kew229. Epub 2016 Jun 21. PMID 27330166
- [Derived] Behrens F, Koehm M, Arndt U, Wittig BM, Greger G, Thaci D, Scharbatke E, Tony HP, Burkhardt H. Does Concomitant Methotrexate with Adalimumab Influence Treatment Outcomes in Patients with Psoriatic Arthritis? Data from a Large Observational Study. J Rheumatol. 2016 Mar;43(3):632-9. doi: 10.3899/jrheum.141596. Epub 2015 Dec 15. PMID 26669916
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psoriatic Arthritis
Started | 4635
Completed | 3569
Not Completed | 1066
Not completed — Adverse Event | 190
Not completed — Lack of Efficacy | 545
Not completed — Lack of Efficacy and Adverse Event | 19
Not completed — Other | 312

BASELINE CHARACTERISTICS:
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 4635
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.4 (11.8)
Gender [Number; unit: participants] — NOTE: gender data were not available for all safety participants
  participants
    Female | 2282
    Male | 2297

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Disease Activity Score (DAS)28
Description: The DAS28 is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, C-reactive protein, and general health are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score greater than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Months 3, 6, 9, 12, 18, and 24
Population: Effectiveness analyses were performed on the full analysis set (FAS). Participants with inadequate data or who met other exclusion criteria were not included in the FAS.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
score on a scale
  Month 3 [N=2757] | -1.7 (1.4)
  Month 6 [N=2412] | -1.9 (1.5)
  Month 9 [N=2028] | -1.9 (1.5)
  Month 12 [N=1850] | -2.0 (1.5)
  Month 18 [N=1572] | -2.0 (1.5)
  Month 24 [N=1315] | -2.1 (1.6)

2. Primary Outcome: Mean Tender Joint Count (TJC) Over Time
Description: Tender joint count represents the number of joints displaying tenderness. Although the DAS28 includes assessments of 28 joints, additional joints are typically evaluated in examinations of participants with Psoriatic Arthritis (PsA) as the joints typically affected in these participants differ from those commonly involved in Rheumatoid Arthritis (RA). Specifically, PsA often involves distal interphalangeal joints (DIP), whereas RA does not.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Tender joints
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
Tender joints
  Baseline [N=3552] | 15.0 (15.3)
  Month 3 [N=3411] | 7.5 (12.3)
  Month 6 [N=2975] | 6.1 (11.3)
  Month 9 [N=2592] | 5.5 (10.9)
  Month 12 [N=2296] | 5.2 (10.5)
  Month 18 [N=1953] | 5.2 (10.5)
  Month 24 [N-1624] | 4.9 (10.4)

3. Primary Outcome: Mean Swollen Joint Count (SJC) Over Time
Description: Swollen joint count represents the number of joints displaying swelling. Although the DAS28 includes assessments of 28 joints, additional joints are typically evaluated in examinations of participants with Psoriatic Arthritis (PsA) as the joints typically affected in these participants differ from those commonly involved in Rheumatoid Arthritis (RA). Specifically, PsA often involves distal interphalangeal joints (DIP), whereas RA does not.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
Swollen Joints
  Baseline [N=3552] | 8.3 (10.2)
  Month 3 [N=3411] | 3.0 (6.9)
  Month 6 [N=2975] | 2.4 (6.3)
  Month 9 [N=2592 | 2.0 (5.5)
  Month 12 [N=2296] | 1.9 (5.6)
  Month 18 [N=1953] | 1.8 (5.2)
  Month 24 [N=1624] | 1.5 (4.5)

4. Primary Outcome: Mean Percent Body Surface Area (BSA) Affected by Psoriasis Over Time
Description: Body surface area was used to evaluate the extent of psoriatic skin involvement. At baseline, investigators classified participants as having BSA less than 3%, 3 to 10%, 11 to 20%, or greater than 20%. At all post-baseline time points, clinicians were asked to estimate BSA on a scale of 0% to 100% rather than as categories. BSA was visually determined by the investigator using the 'rule of nines' and estimating that the palm of the patient's hand was equal to 1% BSA.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
percentage of body surface area
  Baseline [N=3289] | 8.9 (8.4)
  Month 3 [N=2737] | 6.4 (11.2)
  Month 6 [N=2385] | 5.1 (9.7)
  Month 9 [N=2025] | 4.6 (9.9)
  Month 12 [N=1844] | 4.2 (9.3)
  Month 18 [N=1530] | 4.1 (8.9)
  Month 24 [ N=1295] | 4.0 (8.9)

5. Primary Outcome: Mean Target Lesion Score (TLS) Over Time
Description: The Target Lesion Score (TLS) was based on the severity of erythema, scaling, and infiltration of a prospectively-defined psoriasis target lesion of at least 2 cm in width that was considered to be representative of all other affected areas. Each of the three characteristics was evaluated by the clinician on a scale of 0 (absent) to 5 (maximal expression), and these scores were totaled to provide a TLS ranging from 0 (lowest severity) to 15 (highest severity).
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
score on a scale
  Baseline [N=2929] | 6.1 (4.2)
  Month 3 [N=2740] | 3.2 (3.2)
  Month 6 [N=2359] | 2.7 (3.1)
  Month 9 [N=1969] | 2.4 (2.9)
  Month 12 [N=1756] | 2.3 (3.0)
  Month 18 [N=1491] | 2.2 (2.8)
  Month 24 [N=1243] | 2.1 (2.8)

6. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Adverse Events (AEs) were reported that clinicians considered to be related to the study drug. An AE was considered to be a serious adverse event (SAE) if any of the following criteria were met: Death of participant, life-threatening event, hospitalization, prolongation of hospitalization, congenital anomaly, persistent or significant disability or incapacity, important medical event requiring medical or surgical intervention to prevent serious outcome, or spontaneous or elective abortion.
Time Frame: Baseline up to 24 months
Population: Safety Set - All enrolled participants
Measure: Number; unit: participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 4635
participants
  Drug-related AEs excluding SAEs | 877
  SAEs | 143

7. Secondary Outcome: Number of Participants by Severity of Enthesitis Over Time
Description: Enthesitis is a distinguishing characteristic of PsA. Enthesitis involves inflammation at the site where tendons and other connective tissues enter the bone. Investigators reported the presence or absence of enthesitis on the basis of their clinical evaluation; no specific scale or score was used. If present, the severity of each condition was graded by the investigator on a scale of mild, moderate, and severe based on their clinical impression.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
participants
  Baseline, Mild [N=3552] | 422
  Baseline, Moderate [N=3552] | 407
  Baseline, Severe [N=3552] | 119
  Month 3, Mild [N=3432] | 286
  Month 3, Moderate [N=3432] | 130
  Month 3, Severe [N=3432] | 31
  Month 6, Mild [N=2995] | 230
  Month 6, Moderate [N=2995] | 80
  Month 6, Severe [N=2995] | 14
  Month 9, Mild [N=2548] | 188
  Month 9, Moderate [N=2548] | 53
  Month 9, Severe[N=2548] | 12
  Month 12, Mild [N=2307] | 179
  Month 12, Moderate [N=2307] | 46
  Month 12, Severe [N=2307] | 8
  Month 18, Mild [N=1966] | 133
  Month 18, Moderate [N=1966] | 49
  Month 18, Severe [N=1966] | 11
  Month 24, Mild [N=1630] | 107
  Month 24, Moderate [N=1630] | 24
  Month 24, Severe [N=1630] | 5

8. Secondary Outcome: Number of Participants by Severity of Dactylitis Over Time
Description: Dactylitis is a distinguishing characteristic of PsA. Dactylitis, sometimes referred to "sausage digit," involves swelling of the entire finger. Investigators reported the presence or absence of dactylitis on the basis of their clinical evaluation; no specific scale or score was used. If present, the severity of each condition was graded by the investigator on a scale of mild, moderate, and severe based on their clinical impression.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
participants
  Baseline, Mild [N=3552] | 452
  Baseline, Moderate [N=3552] | 765
  Baseline, Severe [N=3552] | 352
  Month 3, Mild [N=3432] | 420
  Month 3, Moderate [N=3432] | 228
  Month 3, Severe [N=3432] | 42
  Month 6, Mild [N=2995] | 313
  Month 6, Moderate [N=2995] | 159
  Month 6, Severe [N=2995] | 23
  Month 9, Mild [N=2548] | 252
  Month 9, Moderate [N=2548] | 114
  Month 9, Severe [N=2548] | 17
  Month 12, Mild [N=2307] | 219
  Month 12, Moderate [N=2307] | 86
  Month 12, Severe [N=2307] | 12
  Month 18, Mild [N=1966] | 167
  Month 18, Moderate [N=1966] | 61
  Month 18, Severe [N=1966] | 8
  Month 24, Mild [N=1630] | 153
  Month 24, Moderate [N=1630] | 41
  Month 24, Severe [N=1630] | 3

9. Secondary Outcome: Number of Participants by Severity of Nail Psoriasis Levels Over Time
Description: Nail psoriasis is a distinguishing characteristic of PsA. Nail psoriasis is characterized by changes in the nail and nail matrix, including pitting, onycholysis (painless separation of the nail from the nail bed), and reddish spots. Investigators reported the presence or absence of nail psoriasis on the basis of their clinical evaluation; no specific scale or score was used. If present, the severity of this condition was graded by the investigator on a scale of mild, moderate, and severe based on their clinical impression.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
participants
  Baseline, Mild [N=3552] | 843
  Baseline, Moderate [N=3552] | 771
  Baseline, Severe [N=3552] | 305
  Month 3, Mild [N=3432] | 996
  Month 3, Moderate [N=3432] | 446
  Month 3, Severe [N=3432] | 99
  Month 6, Mild [N=2995] | 814
  Month 6, Moderate [N=2995] | 266
  Month 6, Severe [N=2995] | 67
  Month 9, Mild [N=2548] | 664
  Month 9, Moderate [N=2548] | 150
  Month 9, Severe [N=2548] | 46
  Month 12, Mild [N=2307] | 595
  Month 12, Moderate [N=2307] | 143
  Month 12, Severe [N=2307] | 30
  Month 18, Mild [N=1966] | 464
  Month 18, Moderate [N=1966] | 123
  Month 18, Severe [N=1966] | 21
  Month 24, Mild [N=1630] | 393
  Month 24, Moderate [N=1630] | 81
  Month 24, Severe [N=1630] | 11

10. Secondary Outcome: Mean Erythrocyte Sedimentation Rate (ESR) Over Time
Description: The Erythrocyte Sedimentation Rate (ESR) is a practicable and sensitive but not specific parameter for measuring disease progression. By means of the ESR it can be generally distinguished between an active and nonactive rheumatic disease. The normal reference range is, as a rule, 0 to 10 mm/h for men and 0 to 15 mm/h for women. The higher the ESR value out of the normal range, the higher is the disease activity.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
mm/hour
  Baseline [N=3149] | 23.3 (20.0)
  Month 3 [N=2925] | 14.3 (14.6)
  Month 6 [N=2566] | 14.2 (14.4)
  Month 9 [N=2161] | 14.3 (14.4)
  Month 12 [N=1970] | 14.5 (14.5)
  Month 18 [N=1659] | 14.5 (13.9)
  Month 24 [N=1391] | 14.5 (13.3)

11. Secondary Outcome: Mean C-Reactive Protein (CRP) Levels Over Time
Description: The C-Reactive Protein (CRP) is an acute phase reactant plasma protein, normally produced by the liver, which is commonly used as an indirect measure of the extent and activity of an inflammation. The CRP normal reference range in the blood is, as a rule, from 0 to 1.0 mg/dL.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
mg/L
  Baseline [N=3522] | 12.8 (26.4)
  Month 3 [N=3022] | 6.2 (12.9)
  Month 6 [N=2642] | 5.9 (10.9)
  Month 9 [N=2247] | 5.6 (10.0)
  Month 12 [N=2047] | 6.0 (18.1)
  Month 18 [N=1751] | 5.4 (10.4)
  Month 24 [N=1440] | 5.4 (23.8)

12. Secondary Outcome: Patients Global Assessment of Disease Activity Over Time
Description: Measured on a visual analog scale (VAS) of 0 to 10 cm; lower scores indicate better participant's status.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
scores on a scale
  Baseline [N=3534] | 6.8 (1.8)
  Month 3 [N=3397] | 3.9 (2.3)
  Month 6 [N=2973] | 3.4 (2.4)
  Month 9 [N=2520] | 3.2 (2.3)
  Month 12 [N=2289] | 3.1 (2.2)
  Month 18 [N=1952] | 3.1 (2.3)
  Month 24 [N=1624] | 2.9 (2.2)

13. Secondary Outcome: Participants Assessment of Fatigue Over Time
Description: Measured on a visual analog scale (VAS) of 0 to 10 cm; lower scores indicate better participant's status.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
scores on a scale
  Baseline [N=3385] | 5.5 (2.7)
  Month 3 [N=3250] | 4.1 (2.7)
  Month 6 [N=2829] | 3.9 (2.7)
  Month 9 [N=2435] | 3.7 (2.7)
  Month 12 [N=2200] | 3.6 (2.6)
  Month 18 [N=1897] | 3.6 (2.7)
  Month 24 [N=1570] | 3.4 (2.6)

14. Secondary Outcome: Participants Assessment of Pain Over Time
Description: Measured on a visual analog scale (VAS) of 0 to 10 cm; lower scores indicate better participant's status.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
scores on a scale
  Baseline [N=3387] | 6.1 (2.2)
  Month 3 [N=3249] | 4.0 (2.5)
  Month 6 [N=2827] | 3.7 (2.5)
  Month 9 [N=2436] | 3.6 (2.5)
  Month 12 [N=2204] | 3.5 (2.5)
  Month 18 [N=1897] | 3.5 (2.6)
  Month 24 [N=1573] | 3.3 (2.4)

15. Secondary Outcome: Mean Funktionsfragebogen Hannover (FFbH) Questionnaire Scores Over Time
Description: A self-administered participant questionnaire used to assess patient function on a scale of 0 (total loss of functional capacity) to 100 (maximal functional capacity) units; the FFbH score indicates the remaining percentage of participant function.
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
scores on a scale
  Baseline [N=3401] | 69.6 (21.1)
  Month 3 [N=3257] | 76.3 (20.7)
  Month 6 [N=2835] | 77.3 (20.9)
  Month 9 [N=2431] | 78.3 (20.8)
  Month 12 [N=2213] | 78.7 (21.1)
  Month 18 [N=1897] | 79.1 (20.8)
  Month 24 [N=1580] | 79.8 (20.5)

16. Secondary Outcome: Percentage of Participants With Impairment in Daily Activities During the Last 4 Weeks of Each Visit
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
percentage of participants
  Baseline, 0 days [N=3307] | 29.3
  Baseline, <7 days [N=3307] | 28.2
  Baseline, 7 to 14 days [N=3307] | 21.7
  Baseline, >14 days [N=3307] | 20.9
  Month 3, 0 days [N=3193] | 49.0
  Month 3, <7 days [N=3193] | 28.4
  Month 3, 7 to 14 days [N=3193] | 13.4
  Month 3, >14 days [N=3193] | 9.2
  Month 6, 0 days [N=2779] | 55.4
  Month 6, <7 days [N=2779] | 25.2
  Month 6, 7 to 14 days [N=2779] | 11.3
  Month 6, >14 days [N=2779] | 8.2
  Month 9, 0 days [N=2390] | 58.5
  Month 9, <7 days [N=2390] | 23.3
  Month 9, 7 to 14 days [N=2390] | 10.6
  Month 9, >14 days [N=2390] | 7.5
  Month 12, 0 days [N=2164] | 59.8
  Month 12, <7 days [N=2164] | 24.2
  Month 12, 7 to 14 days [N=2164] | 9.7
  Month 12, >14 days [N=2164] | 6.4
  Month 18, 0 days [N=1856] | 59.9
  Month 18, <7 days [N=1856] | 25.0
  Month 18, 7 to 14 days [N=1856] | 9.1
  Month 18, >14 days [N=1856] | 6.0
  Month 24, 0 days [N=1553] | 61.6
  Month 24, <7 days [N=1553] | 24.5
  Month 24, 7 to 14 days [N=1553] | 8.6
  Month 24, >14 days [N=1553] | 5.2

17. Secondary Outcome: Mean Number of Days Missed From Work Due to Psoriatic Arthritis
Description: Mean number of days missed from work were derived from patient recall of events in the preceding 12 months (at baseline), in the preceding 3 months (at months 3, 6, 9, and 12), or in the preceding 6 months (at months 18 and 24).
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
days
  Basline [N=2004] | 22.6 (58.2)
  Month 3 [N=1886] | 5.1 (15.7)
  Month 6 [N=1682] | 3.8 (13.5)
  Month 9 [N=1440] | 3.0 (12.5)
  Month 12 [N=1325] | 2.5 (11.2)
  Month 18 [N=1133] | 3.4 (17.9)
  Month 24 [N=929] | 2.8 (16.9)

18. Secondary Outcome: Percentage of Participants With In-Patient Hospitalization
Description: Percentage of participants with in-patient hospitalization were derived from patient recall of events in the preceding 12 months (at Baseline), in the preceding 3 months (at months 3, 6, 9, and 12), or in the preceding 6 months (at months 18 and 24).
Time Frame: Baseline, and Months 3, 6, 9, 12, 18, and 24
Population: as for outcome 1
Measure: Number; unit: percentage of particpants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
percentage of particpants
  Baseline [N=3365] | 17.7
  Month 3 [ N=3232] | 12.0
  Month 6 [N=2804] | 9.1
  Month 9 [N=2417] | 7.0
  Month 12 [N=2183] | 4.8
  Month 18 [N=1877] | 3.8
  Month 24 [N=1568] | 3.3

19. Secondary Outcome: Percentage of Participants on Concomitant Systemic Rheumatic and Pain Relief Medication
Description: Prior and concomitant non-biologic disease-modifying antirheumatic drugs (DMARDs): methotrexate (MTX) and other DMARDs
Time Frame: Baseline, and Months 6 and 24
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 3552
percentage of participants
  Baseline, MTX [N=3552] | 43.7
  Month 6, MTX [N=2823] | 43.2
  Month 24, MTX [N=1555] | 42.7
  Baseline, Other DMARD [N=3552] | 2.4
  Month 6, Other DMARD [N=2823] | 1.4
  Month 24, Other DMARD [N=1555] | 0.9

ADVERSE EVENTS:
Time Frame: From baseline up to 24 months
Description: Other Adverse Events (not including Serious Adverse Events) were measured at >1% frequency, but none occurred above this threshold, therefore 0 is listed for this field.
Arm/Group | Psoriatic Arthritis
Serious Adverse Events (participants affected / at risk) | 143/4635
Other Adverse Events (participants affected / at risk) | 0/4635
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Psoriatic Arthritis (N=4635)
Pneumonia (Infections and infestations) | 7
Erysipelas (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 3
Diverticulitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Acute tonsillitis (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis klebsiella (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Mycotoxicosis (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Skin bacterial infection (Infections and infestations) | 1
Superinfection bacterial (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Appendectomy (Surgical and medical procedures) | 2
Carpal tunnel decompression (Surgical and medical procedures) | 2
Cholecystectomy (Surgical and medical procedures) | 2
Hip arthroplasty (Surgical and medical procedures) | 2
Adhesiolysis (Surgical and medical procedures) | 1
Analgesic therapy (Surgical and medical procedures) | 1
Antibiotics prophylaxis (Surgical and medical procedures) | 1
Aortic bypass (Surgical and medical procedures) | 1
Arthrodesis (Surgical and medical procedures) | 1
Bile duct stent insertion (Surgical and medical procedures) | 1
Breast operation (Surgical and medical procedures) | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 1
Dupuytren's contracture operation (Surgical and medical procedures) | 1
Foot operation (Surgical and medical procedures) | 1
Gallbladder operation (Surgical and medical procedures) | 1
Hospitalization (Surgical and medical procedures) | 1
Hysterectomy (Surgical and medical procedures) | 1
Implantable defibrillator insertion (Surgical and medical procedures) | 1
Intervertebral disc operation (Surgical and medical procedures) | 1
Joint arthroplasty (Surgical and medical procedures) | 1
Knee arthroplasty (Surgical and medical procedures) | 1
Knee operation (Surgical and medical procedures) | 1
Large intestine operation (Surgical and medical procedures) | 1
Lung cyst removal (Surgical and medical procedures) | 1
Osteosynthesis (Surgical and medical procedures) | 1
Percutaneous coronary intervention (Surgical and medical procedures) | 1
Pilonidal sinus repair (Surgical and medical procedures) | 1
Renal stone removal (Surgical and medical procedures) | 1
Shoulder operation (Surgical and medical procedures) | 1
Spinal operation (Surgical and medical procedures) | 1
Stent placement (Surgical and medical procedures) | 1
Thyroid operation (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Ureteral stent insertion (Surgical and medical procedures) | 1
Ureteric calculus removal (Surgical and medical procedures) | 1
Uterine operation (Surgical and medical procedures) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 2
Convulsion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Movement disorder (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Polyneuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pyrexia (General disorders) | 3
Drug ineffective (General disorders) | 2
Cardiac death (General disorders) | 1
Fatigue (General disorders) | 1
Feeling hot (General disorders) | 1
Impaired healing (General disorders) | 1
Injection site urticaria (General disorders) | 1
Malaise (General disorders) | 1
Obstruction (General disorders) | 1
Edema (General disorders) | 1
Edema peripheral (General disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 2
Acute coronary syndrome (Cardiac disorders) | 1
Acute right ventricular failure (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Endocardial disease (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Large intestine perforation (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Lip edema (Gastrointestinal disorders) | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
C-reactive protein increased (Investigations) | 2
Antiphospholipid antibodies positive (Investigations) | 1
Arthroscopy (Investigations) | 1
Biopsy liver (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Body temperature (Investigations) | 1
General physical condition abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Immunology test (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Ureteroscopy (Investigations) | 1
Renal colic (Renal and urinary disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Calculus urinary (Renal and urinary disorders) | 1
Cystitis noninfective (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Traumatic hematoma (Injury, poisoning and procedural complications) | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1
Vasculitis (Vascular disorders) | 2
Circulatory collapse (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Temporal arteritis (Vascular disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Splenic infarction (Blood and lymphatic system disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Hepatocellular damage (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 1
Depression (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Genital rash (Reproductive system and breast disorders) | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Acute vestibular syndrome (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Eyelid edema (Eye disorders) | 1
Walking disability (Social circumstances) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.